CLINICAL TRIAL: NCT05653232
Title: Prophylaxis With Direct-acting Antivirals for Kidney Transplantation From Hepatitis C Virus-Infected Donors to Uninfected Recipients: a Randomized Controlled Trial
Brief Title: Prophylaxis With Direct-acting Antivirals for Kidney Transplantation From HCV-Infected Donors to Uninfected Recipients
Acronym: PREVENT-HCV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00316833; U01AI157931 (NIH)
Record Dates: First submitted 2022-12-06; First posted 2022-12-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: HCV
MeSH Terms: interventions — Disease Transmission, Infectious; Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylaxis (P2W) (Experimental): Prophylaxis is one dose of sofosbuvir/velpatasvir (SOF/VEL) pre-HCV D+/R- kidney transplant (KT), continued for 2 weeks.
  Interventions: Other: Prophylaxis (P2W)
- Transmit and Treat (T&T) (Experimental): T&T is study-supplied SOF/VEL for 12 weeks starting on post-HCV D+/R- kidney transplant day participant's insurance approves standard of care DAAs, or post-KT day 14, whichever comes first.
  Interventions: Other: Transmit and Treat (T&T)

INTERVENTIONS:
Other: Prophylaxis (P2W) — For participants enrolled in P2W arm, the initial dose of SOF/VEL will be administered to the recipient when called to the operating room for transplant (typically 1-3 hours prior to the start of surgery). Post-transplant, SOF/VEL will be continued daily for 13 days post-KT (a total of 14 doses administered).
  Arms: Prophylaxis (P2W)
Other: Transmit and Treat (T&T) — For participants enrolled in T&T arm, SOF/VEL will begin between post-KT day 0 and post-KT day 14. Participants will be clinically-prescribed DAAs once viremia is detected, and participant's insurance will be petitioned to obtain treatment as soon as possible. If insurance-provided DAAs are approved before post-KT day 14, participant will begin 12 weeks of study-provided SOF/VEL on date of insurance-provided DAAs approval. If insurance-provided DAAs are not approved by post-KT day 14, study-provided SOF/VEL will begin on post-KT day 14 and continue for 12 weeks.
  Arms: Transmit and Treat (T&T)

SUMMARY:
This study is being done to find out the best time to start medication for Hepatitis C Virus (HCV) in HCV-negative recipients of HCV-positive (HCV D+/R-) kidney transplants. Participants will be randomized into one of two groups:

Arm 1 - Prophylaxis: This group will start the HCV medication before transplant and will take a shorter course of HCV medication for 2 weeks.

Arm 2 - Transmit and Treat: This group will start the HCV medication after transplant and will take the full course (12 weeks) of HCV medication.

DETAILED DESCRIPTION:
In the past, HCV-positive (HCV+) kidneys were not given to HCV-negative recipients. But over the last few years, medications have been created that cure HCV in nearly 100% of patients. HCV+ transplants to HCV-negative recipients have become increasingly common now that HCV can be cured.

There are two approaches to giving HCV medication to recipients of these transplants. The first is a prophylaxis approach. With prophylaxis, HCV medication is started before transplant and continued for a shorter course after transplant. The second is a transmit-and-treat approach. With transmit-and-treat, HCV medication is started after transplant and continued for the full, recommended course. Both approaches have successfully cured HCV in HCV-negative recipients of HCV+ organs.

This research will use a study drug called sofosbuvir/velpatasvir (SOF/VEL). It contains two drugs for treating HCV in one pill. We will compare giving SOF/VEL for 2 weeks starting pre-transplant (prophylaxis) to giving SOF/VEL for 12 weeks starting no later than 14 days post-transplant (transmit-and-treat).

SOF/VEL belongs to a group of medications called direct-acting antiviral agents (DAAs). These drugs prevent HCV from multiplying and spreading in the human body. SOF/VEL are already approved and used for 12 weeks to treat HCV infection. The use of SOF/VEL for 2 weeks in preventing HCV infection has not been studied. The FDA is allowing SOF/VEL to be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the standard criteria for KT at local center.
* Participant is able to understand and provide informed consent.
* Participant is ≥ 18 years old.

Exclusion Criteria:

* Participant has active HCV infection (detectable HCV RNA) at time of screening.
* Participant has cirrhosis or advanced liver fibrosis.
* Participant's aspartate aminotransferase (AST) or ALT > 2.5 times the upper limit of normal (ULN), within 60 days of screen.
* Participant has human immunodeficiency virus infection (HIV), or active hepatitis B (HBV) infection.
* Participant is unable to safely substitute or discontinue a medication that is contraindicated with the study medication.
* Past or current medical problems, which may pose additional risks from participation in the study, interfere with the participant's ability to comply with study, or impact the quality of the data obtained from the study.
* Participant is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Composite event of HCV-related or HCV treatment-related death, fibrosing cholestatic hepatitis, or HCV relapse | Within 26 weeks of transplant
  Proportion of events in each arm.
Number of participants with liver injury | The first 28 days post-transplant
  Measured with a longitudinal model of Alanine aminotransferase (ALT).

SECONDARY OUTCOMES:
Participant survival | At 6 months and 1 year post-transplant
  Time to event (death)
Graft survival | At 6 months and 1 year post-transplant
  Time to event (graft loss)
HCV plasma RNA | At week 26 post-transplant
  Based on local testing
Graft rejection | At 6 months and 1 year post-transplant
  Cumulative incidence of rejection
Prevalence of donor specific antibody (DSA) | At 4 weeks and 6 months post-transplant, and with any episode of clinically suspected or proven rejection.
  Proportion of participants with a de novo donor-specific human leukocyte antigen (HLA) antibody as measured and reported by local sites' lab
Graft function - eGFR <60 | Months 3, 6, 9, and 12 post-transplant
  Proportion of participants with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - mean eGFR | Months 3, 6, 9, and 12 post-transplant
  Mean calculated eGFR by CKD-EPI
Graft function - eGFR slope | Months 3, 6, 9, and 12 post-transplant
  The slope of eGFR by CKD-EPI, over time based on serum creatinine
Development of HCV resistance-associated variants (RAVs) | With any HCV viremia after P2W or T&T through end of follow up (at least 6 months, up to 3 years post-transplant)
  Proportion of participants with RAVs as measured and reported by local sites' lab
Incidence and severity of bacterial, fungal, viral, and opportunistic infections | From transplant through end of follow up (at least 6 months, up to 3 years post-transplant)
  Cumulative incidence of infections
Incidence of surgical and vascular complications | During the first year post-transplant
  Number of surgical and vascular complications

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - University of California San Diego, La Jolla, California
  - Johns Hopkins University, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Utah Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No